CLINICAL TRIAL: NCT00406211
Title: Follow-up to Evaluate the the Immunogenicity & Safety of GSK Biologicals' MMRV Vaccine Given as a Two-dose Schedule in the Second Year of Life, as Compared to Separate Administration of GSK Biologicals' Priorix® & Varilrix®.
Brief Title: Long-term Follow-up on Immunogenicity & Safety of Measles-Mumps-Rubella-Varicella (MMRV) Combined Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208136/039; 208136/040; 208136/041
Record Dates: First submitted 2006-12-01; First posted 2006-12-04 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Rubella; Varicella; Mumps; Measles
Keywords: Rubella; Varicella; Measles; Mumps; Germany; Austria
MeSH Terms: conditions — Rubella; Chickenpox; Mumps; Measles | interventions — Measles-Mumps-Rubella Vaccine

INTERVENTIONS:
Biological: MMRV
Biological: MMR (Priorix®)
Biological: Varicella (Varilrix®)

SUMMARY:
Follow-up to evaluate the immunogenicity and safety of three production lots of GSK Biologicals' MMRV vaccine given as a two-dose schedule to healthy children in their second year of life, as compared to separate administration of GSK Biologicals' measles-mumps-rubella (MMR) vaccine (Priorix®) and varicella vaccine (Varilrix®) in Germany & Austria. Blood samples were collected at three time points during the follow-up period (Year 1, 2 & 3). No new subjects will be enrolled in these follow-up phases of the study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the parents/guardians of the child before participating in the long-term follow-up.
* Subjects must have received their complete vaccination course according to the group allocation (i.e. subjects must have received either two doses of MMRV combined vaccine, or two doses of Priorix vaccine and one dose of Varilrix vaccine as separate injections in the primary vaccination study.
* Subjects were aged between 12 to 18 months of age at the time of the first vaccination in the primary study.

Exclusion Criteria:

* Subjects must not have received an additional dose of measles, mumps, rubella or varicella containing vaccines.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 398 (Actual)
Dates: Start 2004-07; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Seropositivity rate & antibody titers for MMRV at 1, 2 & 3 year
Occurrence of breakthrough cases & contacts with MMRV disease(s) for 3 years after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (39):
- Austria (4):
  - GSK Investigational Site, Klagenfurt
  - GSK Investigational Site, Neufeld/Leitha
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Villach
- Germany (35):
  - GSK Investigational Site, Bindlach, Bavaria
  - GSK Investigational Site, Marktredwitz, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Tegernsee, Bavaria
  - GSK Investigational Site, Tutzing, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Bad Camberg, Hesse
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Hochheim am Main, Hesse
  - GSK Investigational Site, Marburg/Lahn, Hesse
  - GSK Investigational Site, Nidderau, Hesse
  - GSK Investigational Site, Rüsselsheim am Main, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Salzgitter, Lower Saxony
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Gütersloh, North Rhine-Westphalia
  - GSK Investigational Site, Kirchlengern, North Rhine-Westphalia
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Bad Kreuznach, Rhineland-Palatinate
  - GSK Investigational Site, Bad Sobernheim, Rhineland-Palatinate
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Gau-Algesheim, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Schoeneberg - Kuebelberg, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Worms, Rhineland-Palatinate
  - GSK Investigational Site, Altenholz, Schleswig-Holstein
  - GSK Investigational Site, Bredstedt, Schleswig-Holstein
  - GSK Investigational Site, Brunsbüttel, Schleswig-Holstein
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Husum, Schleswig-Holstein
  - GSK Investigational Site, Neumünster, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Habermehl P, Zepp F, Sänger R, Otto W, Helm K, Meister N, Knuf M, Kindler K, Willems P. Assessment of Varicella Breakthrough Cases One Year after Administration of Two Doses of a Measles, Mumps, Rubella, Varicella Vaccine in the Second Year of Life. Abstract presented at the 24th Annual Meeting of the European Society for Paediatric Infectious Diseases (ESPID), Basel, Switzerland, 03-05 May 2006.
- [Background] Knuf M, Faber J, Barth I, Habermehl P. A combination vaccine against measles, mumps, rubella and varicella. Drugs Today (Barc). 2008 Apr;44(4):279-92. doi: 10.1358/dot.2008.44.4.1210755. PMID 18536786
- [Background] Knuf M, Zepp F, Helm K, Maurer H, Prieler A, Kieninger-Baum D, Douha M, Willems P. Antibody persistence for 3 years following two doses of tetravalent measles-mumps-rubella-varicella vaccine in healthy children. Eur J Pediatr. 2012 Mar;171(3):463-70. doi: 10.1007/s00431-011-1569-4. Epub 2011 Sep 21. PMID 21935584
- [Background] Zepp F et al. Persistence of Functional Antibodies against Mumps Remains High One Year after Administration of Two Doses of a Measles, Mumps, Rubella, Varicella (MMRV) Vaccine in the Second Year of Life. Presented at 24th Annual Meeting of the European Society for Paediatric Infectious Diseases (ESPID), Basel, Switzerland, 03-05 May 2006.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 208136/039 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 208136/039 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 208136/039 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 208136/039 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 208136/039 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 208136/039 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register